CLINICAL TRIAL: NCT00194428
Title: Weight and Metabolic Effects of an Almond Enriched Hypocaloric, Low Fat Diet on Overweight and Obese Persons
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Almond Board of California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 802132
Record Dates: First submitted 2005-09-14; First posted 2005-09-19 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2008-01

CONDITIONS: Obesity; Metabolic Syndrome X; Hyperlipidemia; Hypertension
Keywords: Obesity,; Metabolic Syndrome,; BMI
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Hyperlipidemias; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Almond enriched diet
  Interventions: Behavioral: Almond enriched diet
- 2 (Active Comparator): Low-fat diet
  Interventions: Behavioral: Low fat caloric diet

INTERVENTIONS:
Behavioral: Almond enriched diet — Subjects will consume 2 oz. of almond per day in addition to a low-fat diet
  Other Names: AED
  Arms: 1
Behavioral: Low fat caloric diet — Low fat caloric diet
  Other Names: LFD
  Arms: 2

SUMMARY:
The purpose of this trial is to study the safety, tolerability and efficacy of an almond enriched hypocaloric diet on weight loss and weight maintenance, as well as on established and emerging cardiovascular risk factors in approximately 112 overweight and obese persons.

DETAILED DESCRIPTION:
A randomized, non-blinded, controlled clinical trial using a parallel design of a hypocaloric, low fat (<30% energy from fat) diet with or without 2 oz of almonds over 18 months. Interim analyses will be conducted at 3, 6, 9 and 12 months. The study will be divided into 3 phases. Phase 1 (months 0-6) will be an active, intensive weight loss phase. During phase 1, all subjects will meet once a week in the evening for 1.5 hours. Phase 2 (months 6-12) will be a less intensive weight loss phase. During phase 2 groups will meet every other week in the evening for 1.5 hours. The last phase will be the weight maintenance phase or phase 3 (months 12-18).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) > 27 but <40
* 18-75 years of age
* Men and non-pregnant or lactating women
* Subjects must be willing to comply with all study-related procedures

Exclusion Criteria:

* Uncontrolled hypertension
* Diabetes or use of anti-hyperglycemic medication
* Dyslipidemia requiring prescription drug therapy as defined by NCEP ATPIII guidelines at screening
* Known allergy or sensitivity to nuts
* Known atherosclerotic cardiovascular disease
* History of congestive heart failure
* History of a non-skin malignancy within the previous 5 years
* Any major active rheumatologic, pulmonary, hepatic, renal, dermatologic disease or inflammatory condition
* History of being HIV positive
* History of alcohol or drug abuse
* Weight-loss inducing medications or dietary supplements within 3 months prior to enrollment.
* Weight loss > 5 kg during the last 6 months
* Participation in an investigational drug study within 6 weeks prior to screening
* Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2005-02; Primary Completion 2007-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of an almond-enriched (2 oz/day) hypocaloric, low-fat diet on body weight and body composition in overweight and obese persons | 6 months

SECONDARY OUTCOMES:
To evaluate the effects of the almond enriched diet on established and emerging surrogate markers of coronoary artery disease (CAD) risk | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gary D Foster, PhD, Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Jenkins DJ, Kendall CW, Marchie A, Faulkner D, Vidgen E, Lapsley KG, Trautwein EA, Parker TL, Josse RG, Leiter LA, Connelly PW. The effect of combining plant sterols, soy protein, viscous fibers, and almonds in treating hypercholesterolemia. Metabolism. 2003 Nov;52(11):1478-83. doi: 10.1016/s0026-0495(03)00260-9. PMID 14624410
- [Background] Wien MA, Sabate JM, Ikle DN, Cole SE, Kandeel FR. Almonds vs complex carbohydrates in a weight reduction program. Int J Obes Relat Metab Disord. 2003 Nov;27(11):1365-72. doi: 10.1038/sj.ijo.0802411. PMID 14574348
- [Derived] Foster GD, Shantz KL, Vander Veur SS, Oliver TL, Lent MR, Virus A, Szapary PO, Rader DJ, Zemel BS, Gilden-Tsai A. A randomized trial of the effects of an almond-enriched, hypocaloric diet in the treatment of obesity. Am J Clin Nutr. 2012 Aug;96(2):249-54. doi: 10.3945/ajcn.112.037895. Epub 2012 Jun 27. PMID 22743313
- See also: Related Info — http://www.almondsarein.com
- See also: Related Info — http://www.almondboard.com